CLINICAL TRIAL: NCT00425529
Title: Tolerance and Practicality of Module AOX - a Modular Device for Supplementation of Enteral Nutrition
Brief Title: Tolerance and Practicality of Module AOX
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 01.04.CLI
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2007-01-23 (Estimated); Status verified 2007-01

CONDITIONS: Gastrointestinal Diseases; Nutrition
MeSH Terms: conditions — Gastrointestinal Diseases

INTERVENTIONS:
Device: Module AOX (attached to Sondalis ISO)

SUMMARY:
The primary objective of this clinical trial is to test the tolerance and practicality of the new device Module AOX.

The secondary objective is to determine the changes in oxidative, antioxidative status, plasma free amino acids, and various immune parameters in critically ill patients receiving the enteral nutrition with and without using Module AOX.

DETAILED DESCRIPTION:
Surgery and trauma induce hypercatabolism accompanied by a systemic immunoinflammtory response and massive production of reactive oxygen species at the site of injury. In these situations, requirements for certain amino acids (glutamine, cysteine) and antioxidant micronutrients (zinc, vitamin E, vitamin C, beta-caroteen, selenium) are markedly increased and may not be covered by the levels normally present in standard enteral diets, especially in the early phase when enteral nutrition is introduced gradually. Thus, supplementation with amino acids and antioxidant micronutrients may be appropiate in order to optimize nutritional support in such patients.

The administration of selected nutrients via modular devices added to a standard enteral formulation is an attractive means of providing optimized nutrition support for specific disease states. Module AOX is intended for supplementation of patients requiring nutritional support for a condition in which oxidative stress is expected. The module contains:

* Glutamine: to support gut mucosal and immune function, to minimize early depletion of glutamine stores and preserve body protein
* Cysteine: to support synthesis of glutathione, an important cellular antioxidant, and to support the synthesis of acute phase proteins
* Vitamin E, vitamin C and beta-caroteen: water- and lipid-soluble antioxidant micronutrients to boost antioxidant defenses
* Zinc: to compensate for increased losses and to support protein synthesis, immune function and wound healing
* Selenium: to compensate for increased losses, support antioxidant defenses and immune function

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo major surgery of esophagus, stomach or pancreas
* patients who will be eligible for jejunostomy feeding
* age >18 and <75 y
* BMI < 35
* having obtained his/her or his/her legal representative's informed consent

Exclusion Criteria:

* patients with a history of main cardiovascular or kidney disease
* weigth loss >10% during the last 6 months
* patients who have received corticosteroids, or investigational drugs, in the last 6 weekd prior to surgery
* patients with HIV infection
* patients who are participating in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-02; Study Completion 2003-05

PRIMARY OUTCOMES:
Tolerance: stool outcome (frequency, consistency), diarrhea, faltulence, abdominal pain, amount of feeding according to goal, changes of amount fed, discontinuation of feeding
Practicality: time for connecting the device to the pouch, time needing for mixing content of device with the content of the enteral feding pouch, clotting of theadministration set, product flow,leakage, clarity of instructions of usage

SECONDARY OUTCOMES:
vitamin C, Vitamin E. beta-caroteen, GSH/GSSG, cysteine/cystine, GPx, isoprostane, TAS, Zn, Se, plasma free amino acids, HLADR, TNF soluble receptors (55/75), LBP, BPI, IL-1 IR II, leptin, soluble leptin receptor, IL-6, IL-8, and microciological safety

CONTACTS AND LOCATIONS:
Overall Officials: Paul AM van Leeuwen, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands